CLINICAL TRIAL: NCT00381615
Title: A Phase 2, Open Label, Multi-Center, Controlled, Randomized Study of the Safety, Tolerability and Immunogenicity of Novartis Meningococcal B Recombinant Vaccine±OMV, When Administered to Healthy Infants at 2, 4, 6 and/or 12 Months of Age
Brief Title: Prevention, Randomized, Open Label, Active Control, Parallel Assignment, Safety/Efficacy Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72P6
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Meningococcal disease; prevention; vaccination
MeSH Terms: conditions — Meningococcal Infections | interventions — diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; Tetanus Toxoid; Poliovirus Vaccine, Inactivated; Heptavalent Pneumococcal Conjugate Vaccine; MenC-CRM vaccine; Rubella Vaccine; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- rMenB (Experimental): Infants received 4 doses of recombinant meningococcal serogroup B (rMenB) vaccine without outer membrane vesicle (OMV-NZ) at 2, 4, 6 and 12 months of age.
  Infants also received routine vaccines - 3 doses each of Diphtheria Tetanus Pertussis-Haemophilus influenzae type b-Inactivated Polio Vaccine (DTaP-Hib-IPV) (at 2, 3, and 4 months) and Heptavalent Pneumococcal Conjugate (PC7) (at 2, 4 and 13 months), 2 doses of MenC-CRM (at 3 and 5 months) and 1 dose each of MenC-Hib (at 12 months) and Measles Mumps Rubella (MMR) (at 13 months).
  Interventions: Biological: rMenB; Biological: DTaP-Hib-IPV; Biological: PC7; Biological: MenC-CRM; Biological: MenC-Hib; Biological: MMR
- rMenB+OMV (Experimental): Infants received 4 doses of rMenB vaccine with OMV-NZ at 2, 4, 6 and 12 months of age.
  Infants also received routine vaccines - 3 doses each of DTaP-Hib-IPV (at 2, 3, and 4 months) and PC7 (at 2, 4 and 13 months), 2 doses of MenC-CRM (at 3 and 5 months) and 1 dose each of MenC-Hib (at 12 months) and MMR (at 13 months).
  Interventions: Biological: rMenB+OMV; Biological: DTaP-Hib-IPV; Biological: PC7; Biological: MenC-CRM; Biological: MenC-Hib; Biological: MMR
- Routine (Experimental): Infants received routine vaccines - 3 doses each of DTaP-Hib-IPV (at 2, 3, and 4 months) and PC7 (at 2, 4 and 13 months), 2 doses of MenC-CRM (at 3 and 5 months) and 1 dose each of MenC-Hib (at 12 months) and MMR (at 13 months).
  Infants also received single dose of rMenB vaccine without OMV-NZ at 12 months of age.
  Interventions: Biological: rMenB; Biological: DTaP-Hib-IPV; Biological: PC7; Biological: MenC-CRM; Biological: MenC-Hib; Biological: MMR
- Routine+OMV (Experimental): Infants received routine vaccines - 3 doses each of DTaP-Hib-IPV (at 2, 3, and 4 months) and PC7 (at 2, 4 and 13 months), 2 doses of MenC-CRM (at 3 and 5 months) and 1 dose each of MenC-Hib (at 12 months) and MMR (at 13 months).
  Infants also received single dose of rMenB vaccine with OMV-NZ at 12 months of age.
  Interventions: Biological: rMenB+OMV; Biological: DTaP-Hib-IPV; Biological: PC7; Biological: MenC-CRM; Biological: MenC-Hib; Biological: MMR

INTERVENTIONS:
Biological: rMenB — One dose (0.5 mL) of rMenB vaccine without OMV-NZ supplied as a full liquid formulation in a prefilled syringe was administered into the anterolateral area of the right thigh.
  Other Names: Serogroup B meningococcal recombinant vaccine without OMV-NZ
  Arms: Routine; rMenB
Biological: rMenB+OMV — One dose (0.5 mL) of rMenB vaccine with OMV-NZ supplied as a full liquid formulation in a prefilled syringe was administered into the anterolateral area of the right thigh.
  Other Names: Serogroup B meningococcal recombinant vaccine with OMV-NZ
  Arms: Routine+OMV; rMenB+OMV
Biological: DTaP-Hib-IPV — Intramuscular (IM) injections of 3 doses of 0.5 mL each of DTaP-Hib-IPV supplied in prefilled vial were administered at 2, 3 and 4 months in the anterolateral area of the left thigh (when given concomitantly with rMenB±OMV-NZ) or the right thigh.
  Other Names: Combined diphtheria, tetanus toxoid, acellular pertussis, Haemophilus influenzae type B; and inactivated polio vaccine; Pediacel
Biological: PC7 — IM injections of 3 doses of 0.5 mL each of PC7 supplied in prefilled syringe were administered at 2, 4 and 13 months of age in the anterolateral area of the left thigh (when given concomitantly with rMenB±OMV-NZ) or the right thigh.
  Other Names: Heptavalent Streptoccus pneumonia vaccine; Prevenar
Biological: MenC-CRM — MenC-CRM was obtained by extemporaneous mixing just before injection of the lyophilized Men C component to be re-suspended with the saline solvent (aluminum hydroxide suspension) supplied. IM injection of 2 doses each of 0.5 mL were administered into the anterolateral area of the left thigh.
  Other Names: CRM197 conjugated meningococcal C vaccine; Menjugate
Biological: MenC-Hib — MenC-Hib was obtained by extemporaneous mixing of powder and solvent just before injection. One dose (0.5 mL) of MenC-Hib was administered at 12 months of age as an IM injection into the anterolateral area of the thigh.
  Other Names: Combined meningococcal C and Haemophilus influenzae type B vaccine; Menitorix
Biological: MMR — IM injection of one dose of 0.5 mL of MMR obtained by extemporaneous mixing just before injection of powder and the solvent for solution was administered at 13 months of age in the anterolateral area of the left thigh.
  Other Names: Measles, mumps, and rubella vaccine; Priorix

SUMMARY:
This study was aimed to explore safety and immunogenicity of two formulations of a Meningococcal B Vaccine when administered to healthy infants.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible to be enrolled in the study:

1. healthy 2-month old infants (55-89 days, inclusive), born after full term pregnancy with an estimated gestational age ≥37 weeks and a birth weight ≥2.5 kg;
2. for whom a parent/legal guardian had provided written informed consent after the nature of the study had been explained;
3. those available for all the visits scheduled in the study;
4. those in good health as determined by:

   1. medical history
   2. physical examination
   3. clinical judgment of the investigator

Exclusion Criteria:

Individuals were not to be enrolled into the study:

1. whose parents/legal guardians were unwilling or unable to give written informed consent to participate in the study; 2. who had previously received any meningococcal B vaccine; 3. who had received prior vaccination with Diphtheria Tetanus Pertussis (DTP) (acellular or whole cell), Inactivated Polio Vaccine (IPV) or Oral Polio Vaccine (OPV), H influenzae type b (Hib) or Heptavalent Pneumococcal Conjugate (PC7) vaccine; 4. who had a previous ascertained or suspected disease caused by N meningitidis, S pneumoniae, C diphtheriae, tetani, Poliovirus, Hib, or B pertussis (history of laboratory confirmed, or clinical condition of spasmodic cough for a period ≥2weeks associated with apnea or whooping); 5. who had household contact with and/or intimate exposure to an individual with laboratory confirmed N meningitidis, B pertussis, Hib, C diphtheriae or Polio infection since birth; 6. who had a history of any anaphylactic shock, asthma, urticaria or other allergic reaction after previous vaccinations or known hypersensitivity to any vaccine component; 7. who had experienced significant acute or chronic infection within the previous 7 days or had experienced fever (≥38.0°C) within the previous 3 days; 8. who had any present or suspected serious acute or chronic disease (e.g., with signs of cardiac, renal failure, hepatic disease, or severe malnutrition or insulin dependent diabetes), or progressive neurological disease, or a genetic anomaly/known cytogenic disorders (e.g., Down's syndrome); 9. who had leukemia, lymphomas; 10. who had a known or suspected autoimmune disease or impairment/alteration of immune function resulting from (for example):

1. receipt of any immunosuppressive therapy since birth
2. receipt of immunostimulants since birth
3. receipt of any systemic corticosteroid since birth 11. with a suspected or known HIV infection or HIV related disease; 12. who had ever received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation from birth and for the full length of the study; 13. with a known bleeding diathesis, or any condition that might be associated with a prolonged bleeding time; 14. who had experienced any seizure, either associated with fever or as part of an underlying neurological disorder or syndrome 15. who had taken antibiotics within 7 days prior to enrollment (exception: antibiotics taken once daily within 14 days after the last dose); 16. who had either received, or for whom there was intent to immunize with any other vaccine(s), with respect to the study vaccines, within 30 days prior and throughout the study period; 17. who had ever received another investigational agent from birth prior to enrollment and unwilling to refuse participation in another investigational trial through the end of the study; 18. whose parents/legal guardians, were planning to leave the area of the study site before the end of the study period; 19. with any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 55 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Information Services, Study Chair — Novartis
Locations (3):
- United Kingdom (3):
  - Gloucester
  - London
  - Oxford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at three study centers in the United Kingdom (UK).
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- rMenB: Infants received 4 doses of recombinant meningococcal serogroup B (rMenB) vaccine without Outer Membrane Vesicle (OMV-NZ) at 2, 4, 6 and 12 months of age.
  Infants also received routine vaccines - 3 doses each of diphtheria-tetanus-acellular pertussis vaccine (DTaP-Hib-IPV) (at 2, 3, and 4 months) and Heptavalent Pneumococcal Conjugate (PC7) (at 2, 4 and 13 months), 2 doses of MenC-CRM (at 3 and 5 months) and 1 dose each of MenC-Hib (at 12 months) and Measles Mumps Rubella (MMR) (at 13 months).
Period: Overall Study
Arm/Group | rMenB | rMenB+OMV | Routine | Routine+OMV
Started | 48 | 50 | 25 | 24
Completed | 44 | 45 | 24 | 22
Not Completed | 4 | 5 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 1
Not completed — Lost to Follow-up | 3 | 2 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled subjects.
Groups:
- rMenB: Infants received 4 doses of rMenB vaccine without OMV-NZ at 2, 4, 6 and 12 months of age.
  Infants also received routine vaccines - 3 doses each of DTaP-Hib-IPV (at 2, 3, and 4 months) and PC7 (at 2, 4 and 13 months), 2 doses of MenC-CRM (at 3 and 5 months) and 1 dose each of MenC-Hib (at 12 months) and MMR (at 13 months).
- Total: Total of all reporting groups
Arm/Group | rMenB | rMenB+OMV | Routine | Routine+OMV | Total
Number analyzed (Participants) | 48 | 50 | 25 | 24 | 147
Age, Continuous [Mean (Standard Deviation); unit: Days] | 59.0 (3.4) | 60.9 (5.9) | 60.4 (5.9) | 60.9 (6.1) | 60.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 9 | 7 | 62
  Male | 24 | 28 | 16 | 17 | 85

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Bactericidal Titers, BCA ≥1:4, 30 Days After the Third Immunization
Description: Immunogenicity was measured as percentage of subjects who achieved bactericidal titers ≥1:4 against meningococcal strains 44/76-SL, 5/99 and NZ98/254, evaluated using serum bactericidal assay, before vaccination (baseline) and at one month after third-dose of Infants series vaccination of rMenB vaccine with and without OMV administered at 6 months of age.
Time Frame: Baseline and one month after third-dose of infants series
Population: Analysis was performed on the per protocol (PP) set, i.e. all subjects in the enrolled population who received all the relevant doses of vaccine correctly; provided evaluable serum samples at the relevant time points, and had no major protocol violation as defined prior to analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 46 | 46
Percentage of subjects
  Strain 44/76-SL - Titer ≥1:4 - Baseline | 11 [4 to 24] | 11 [4 to 24]
  Str. 44/76-SL-Titer ≥1:4- Post-3rd dose (N=36,39) | 78 [61 to 90] | 87 [73 to 96]
  Strain 5/99 - Titer ≥1:4 - Baseline (N=42,43) | 7 [1 to 19] | 14 [5 to 28]
  Str. 5/99 - Titer ≥1:4- Post-3rd dose (N=32,37) | 100 [89 to 100] | 95 [82 to 99]
  Strain NZ98/254 - Titer ≥1:4 - Baseline (N=46,46) | 4 [1 to 15] | 9 [2 to 21]
  Str. NZ98/254-Titer ≥1:4- Post-3rd dose (N=37,40) | 5 [1 to 18] | 85 [70 to 94]

2. Secondary Outcome: Percentages of Subjects With Fourfold Rises in Bactericidal Titers 1 Month After First Vaccination
Description: Percentages of subjects treated with Routine + Novartis rMenB Vaccine +/- OMV NZ (Groups III and IV) with fourfold rises in bactericidal titers for the three major meningococcal B strains (Strain 44/76-SL, Strain 5/99, Strain NZ98/254) 1 month after first vaccination. The analysis was done on the Per Protocol population 1 month after first vaccination.
Time Frame: 1 month after first vaccination
Population: Analysis was performed on the PP set.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Routine: Infants received routine vaccines - 3 doses each of DTaP-Hib-IPV (at 2, 3, and 4 months) and PC7 (at 2, 4 and 13 months), 2 doses of MenC-CRM (at 3 and 5 months) and 1 dose each of MenC-Hib (at 12 months) and MMR (at 13 months). Infants also received single dose of rMenB vaccine without OMV NZ at 12 months of age.
- Routine+OMV: Infants received routine vaccines - 3 doses each of DTaP-Hib-IPV (at 2, 3, and 4 months) and PC7 (at 2, 4 and 13 months), 2 doses of MenC-CRM (at 3 and 5 months) and 1 dose each of MenC-Hib (at 12 months) and MMR (at 13 months). Infants also received single dose of rMenB vaccine with OMV NZ at 12 months of age.
Arm/Group | Routine | Routine+OMV
Number analyzed (Participants) | 22 | 22
Percentage of subjects
  44/76-SL (1 month after first Vacc; N=22, 22) | 14 [3 to 35] | 36 [17 to 59]
  5/99 (1 month after first Vacc; N=21, 22) | 100 [84 to 100] | 59 [36 to 79]
  NZ98/254 (1 month after first Vacc; N=21, 22) | 0 [0 to 16] | 9 [1 to 29]
  44/76-SL (1 month after 4th (booster); N=37, 30) | 92 [78 to 98] | 93 [78 to 99]
  5/99 (1 month after 4th (booster); N=33, 27) | 97 [85 to 100] | 97 [83 to 100]
  NZ98/254 (1 month after 4th (booster); N=38, 29) | 0 [0 to 9] | 76 [56 to 90]

3. Primary Outcome: Geometric Mean Bactericidal Titers Against Meningococcal Strains One Month After Third-Dose of Infants Series Vaccination of rMenB Vaccine With and Without OMV-NZ
Description: The immune response was measured as the geometric mean bactericidal titers directed against meningococcal strains 44/76-SL, 5/99 and NZ98/254, before vaccination (baseline) and at one month after third-dose of infants series vaccination of rMenB vaccine with and without OMV administered at 6 months of age.
Time Frame: Baseline and one month after third-dose of infants series
Population: Analysis was performed on the PP set.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 46 | 46
titers
  Strain 44/76-SL - Baseline | 1.32 [1.05 to 1.66] | 1.4 [1.16 to 1.69]
  Strain 44/76-SL - Post-3rd dose (N=36,39) | 13 [8.11 to 22] | 30 [19 to 46]
  Strain 5/99 - Baseline (N=42,43) | 1.22 [0.98 to 1.52] | 1.43 [1.12 to 1.81]
  Strain 5/99 - Post-3rd dose (N=32,37) | 159 [100 to 253] | 126 [77 to 205]
  Strain NZ98/254 - Baseline (N=46,46) | 1.23 [1 to 1.52] | 1.15 [1.02 to 1.29]
  Strain NZ98/254 - Post-3rd dose (N=37,40) | 1.16 [0.98 to 1.38] | 19 [11 to 33]

4. Secondary Outcome: Geometric Mean Titers Against a Panel of Genetically Distinct Meningococcal Strains Prior to the First Dose, 30 Days After the Second Immunization and at 12 Months Age
Description: Geometric mean bactericidal titers as measure of the Bactericidal activity against meningococcal strains 44/76-SL, 5/99 and NZ98/254, before vaccination (baseline) and at 30 days after second immunization, at 12 months age,and 30 days after the fourth (booster) vaccination.
Time Frame: prior 1st dose, 30 days post-2nd vaccination, 12 months age to 1 month post 4th vaccination
Population: Analysis was performed on the PP set.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 46 | 46
titers
  Strain 44/76-SL (pre-vaccination; N=45, 45) | 1.32 [1.05 to 1.66] | 1.4 [1.16 to 1.69]
  Strain 5/99 (pre-vaccination; N=42, 43) | 1.22 [0.98 to 1.52] | 1.43 [1.12 to 1.81]
  Strain NZ98/254 (pre-vaccination; N=46, 46) | 1.23 [1 to 1.52] | 1.15 [1.02 to 1.29]
  Strain 44/76-SL (1 Month After 2nd Vacc; N=40, 37) | 5.96 [3.94 to 9.01] | 28 [19 to 40]
  Strain 5/99 (1 Month After 2nd Vacc; N=36, 33) | 119 [63 to 223] | 104 [64 to 169]
  Strain NZ98/254 (1 Month After 2nd Vacc; N=41, 38) | 1.13 [0.97 to 1.31] | 6.55 [4.77 to 8.99]
  44/76-SL (6 months after pre-booster; N=40, 44) | 5.46 [4.06 to 7.35] | 5.07 [3.62 to 7.1]
  5/99 (6 months after pre-booster; N=37, 40) | 37 [23 to 61] | 21 [13 to 37]
  NZ98/254 (6 months after pre-booster; N=41, 44) | 1.14 [0.95 to 1.38] | 2.38 [1.65 to 3.43]
  44/76-SL (1 month after booster; N=38, 31) | 56 [40 to 79] | 114 [76 to 173]
  5/99 (1 month after booster; N=34, 30) | 261 [157 to 435] | 691 [357 to 1340]
  NZ98/254 (1 month after booster; N=39, 31) | 1.09 [0.91 to 1.31] | 33 [17 to 61]

5. Secondary Outcome: Geometric Mean Titers Against a Panel of Genetically Distinct Meningococcal Strains Prior to and 30 Days After a Single Dose Administered at 12 Months of ageVaccination of rMenB Vaccine With and Without OMV-NZ
Description: Geometric Mean Titers (GMTs) as measure of the bactericidal activity against the for the three major meningococcal B strains (Strain 44/76-SL, Strain 5/99, Strain NZ98/254) in subjects treated with Routine +Novartis rMenB Vaccine +/- OMV NZ (Groups III and IV) at 12 months age, i.e. pre-first vaccination and 1 month after first vaccination. The analysis was done on the Per Protocol population.
Time Frame: pre-first vaccination and 1 month after first vaccination
Population: Analysis was performed on the PP set.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Routine | Routine+OMV
Number analyzed (Participants) | 22 | 22
titers
  44/76-SL (pre-vaccination; N=22,22) | 1.55 [1.22 to 1.98] | 1.88 [1.19 to 2.96]
  5/99 (pre-vaccination; N=21,22) | 1 [1 to 1] | 1 [1 to 1]
  NZ98/254 (pre-vaccination; N=21, 22) | 1.03 [0.96 to 1.11] | 1 [1 to 1]
  44/76-SL (1 month after first Vacc; N=22,22) | 2.34 [1.66 to 3.29] | 6.02 [3.5 to 10]
  5/99 (1 month after first Vacc; N=21,22) | 73 [53 to 101] | 8 [4.2 to 15]
  NZ98/254 (1 month after first Vacc; N=21, 22) | 1 [1 to 1] | 1.66 [1.12 to 2.45]

6. Secondary Outcome: Geometric Mean Ratios (GMRs) to Baseline Against a Panel of Genetically Distinct Meningococcal Strains 30 Days After the Second Immunization and 1 Month After Fourth (Booster) Vaccination
Description: Geometric Mean Ratios (GMRs) as measure of the bactericidal activity against meningococcal B strains (Strain 44/76-SL, Strain 5/99, Strain NZ98/254) in subjects treated with Novartis rMenB Vaccine +/- OMV NZ (Groups I and II) at 30 days after the second immunization and 1 month after fourth (booster) vaccination. The analysis was done on the Per Protocol population at 30 days after the second immunization and 1 month after fourth (booster) vaccination.of age.
Time Frame: 30 days after the second vaccination and 1 month after fourth (booster) vaccination
Population: Analysis was performed on the PP set.
Measure: Geometric Mean (95% Confidence Interval); unit: ratios
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 41 | 38
ratios
  Strain 44/76-SL (1 Month After 2nd Vacc; N=40, 37) | 4.36 [2.78 to 6.84] | 19 [13 to 29]
  Strain 5/99 (1 Month After 2nd Vacc; N=36, 33) | 104 [54 to 200] | 71 [44 to 115]
  Strain NZ98/254 (1 Month After 2nd Vacc; N=41, 38) | 0.92 [0.69 to 1.22] | 5.55 [3.9 to 7.92]
  44/76-SL (1 month after booster; N=38, 31) | 42 [28 to 64] | 78 [47 to 130]
  5/99 (1 month after booster; N=34, 30) | 217 [128 to 370] | 467 [231 to 945]
  NZ98/254 (1 month after booster; N=39, 31) | 0.85 [0.62 to 1.16] | 28 [15 to 52]

7. Secondary Outcome: Percentages of Subjects With Bactericidal Titers ≥1:4 at 12 Months Age
Description: Percentages of subjects treated with Routine + Novartis rMenB Vaccine +/- OMV NZ (Groups III and IV) with a bactericidal activity (BCA) measured as BCA titer ≥1:4 for the for three major meningococcal B strains (Strain 44/76-SL, Strain 5/99, Strain NZ98/254) at 12 months age, i.e. pre-first vaccination, and 1 month after first vaccination. The analysis was done on the Per Protocol population at 12 months age, i.e. pre-first vaccination, and 1 month after first vaccination.
Time Frame: pre-first vaccination and 1 month after first vaccination
Population: Analysis was performed on the PP set after booster vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Routine | Routine+OMV
Number analyzed (Participants) | 22 | 22
Percentage of subjects
  44/76-SL (12 Months Age, pre-first vacc; N=22,22) | 9 [1 to 29] | 18 [5 to 40]
  5/99 (12 Months of Age, pre-first vacc; N=21,22) | 0 [0 to 16] | 0 [0 to 15]
  NZ98/254 (12 Months Age, pre-first vacc; N=21,22) | 0 [0 to 16] | 0 [0 to 15]
  44/76-SL (1 month after first Vacc; N=22,22) | 32 [14 to 55] | 73 [50 to 89]
  5/99 (1 month after first Vacc; N=21,22) | 100 [84 to 100] | 73 [50 to 89]
  NZ98/254 (1 month after first Vacc; N=21, 22) | 0 [0 to 16] | 18 [5 to 40]

8. Primary Outcome: Number of Subjects Who Reported Solicited Local Reactions After Each Vaccination of rMenB Vaccine With and Without OMV
Description: Safety was assessed as the number of subjects who reported solicited local reactions from day 1 through day 7 after each vaccination of rMenB vaccine with and without OMV administered at 2 months (vaccination 1), 4 months (vaccination 2), 6 months (vaccination 3) and 12 months (vaccination 4; vaccination 1 for Routine and Routine+OMV groups).
Time Frame: Day 1 through day 7 after each vaccination
Population: Analysis was performed on the safety set, i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: Number of subjects
Arm/Group | rMenB | rMenB+OMV | Routine | Routine+OMV
Number analyzed (Participants) | 48 | 50 | 24 | 23
Number of subjects
  Tenderness - Vaccination 1 | 17 | 17 | 0 | 0
  Tenderness - Vaccination 2 (N=48,48,24,23) | 10 | 14 | 0 | 0
  Tenderness - Vaccination 3 (N=47,48,24,23) | 10 | 17 | 6 | 7
  Tenderness - Vaccination 4 (N=45,48,24,23) | 10 | 23 | 0 | 0
  Erythema - Vaccination 1 | 40 | 42 | 0 | 0
  Erythema - Vaccination 2 (N=48,48,24,23) | 43 | 45 | 0 | 0
  Erythema - Vaccination 3 (N=47,48,24,23) | 43 | 44 | 0 | 0
  Erythema - Vaccination 4 (N=45,48,24,23) | 43 | 46 | 0 | 0
  Induration - Vaccination 1 | 15 | 24 | 0 | 0
  Induration - Vaccination 2 (N=48,48,24,23) | 13 | 24 | 0 | 0
  Induration - Vaccination 3 (N=47,48,24,23) | 20 | 22 | 10 | 19
  Induration - Vaccination 4 (N=45,48,24,23) | 22 | 34 | 0 | 0

9. Primary Outcome: Number of Subjects Who Reported Solicited Local Reactions After Each Vaccination of PC7
Description: Safety was assessed as the number of subjects who reported solicited local reactions from day 1 through day 7 after each vaccination of PC7 administered at 2 months (vaccination 1) and 4 months (vaccination 3).
Time Frame: Day 1 through day 7 after each vaccination
Population: Analysis was performed on the safety set.
Measure: Number; unit: Number of subjects
Arm/Group | rMenB | rMenB+OMV | Routine | Routine+OMV
Number analyzed (Participants) | 48 | 50 | 25 | 24
Number of subjects
  Tenderness - Vaccination 1 | 19 | 21 | 7 | 10
  Tenderness - Vaccination 3 (N=48,48,25,24) | 10 | 12 | 6 | 6
  Erythema - Vaccination 1 | 38 | 43 | 24 | 20
  Erythema - Vaccination 3 (N=48,48,25,24) | 43 | 42 | 24 | 22
  Induration - Vaccination 1 | 19 | 21 | 11 | 13
  Induration - Vaccination 3 (N=48,48,25,24) | 19 | 19 | 13 | 16

10. Primary Outcome: Number of Subjects Who Reported Solicited Local Reactions After Each Vaccination of DTaP-Hib-IPV Pentavalent Vaccine
Description: Safety was assessed as the number of subjects who reported solicited local reactions from day 1 through day 7 after each vaccination of the pentavalent vaccine DTaP-Hib-IPV administered at 2 months (vaccination 1), 3 months (vaccination 2) and 4 months (vaccination 3).
Time Frame: Day 1 through day 7 after each vaccination
Population: Analysis was performed on the safety set.
Measure: Number; unit: Number of subjects
Arm/Group | rMenB | rMenB+OMV | Routine | Routine+OMV
Number analyzed (Participants) | 48 | 50 | 25 | 24
Number of subjects
  Tenderness - Vaccination 1 | 21 | 22 | 8 | 14
  Tenderness - Vaccination 2 (N=48,49,25,24) | 14 | 8 | 5 | 5
  Tenderness - Vaccination 3 (N=48,48,25,24) | 12 | 12 | 3 | 6
  Erythema - Vaccination 1 | 37 | 41 | 24 | 22
  Erythema - Vaccination 2 (N=48,49,25,24) | 42 | 44 | 25 | 22
  Erythema - Vaccination 3 (N=48,48,25,24) | 41 | 42 | 24 | 23
  Induration - Vaccination 1 | 19 | 20 | 10 | 16
  Induration - Vaccination 2 (N=48,49,25,24) | 17 | 16 | 8 | 11
  Induration - Vaccination 3 (N=48,48,25,24) | 23 | 20 | 13 | 15

11. Primary Outcome: Number of Subjects Who Reported Solicited Local Reactions After Each Vaccination of MenC-CRM or MenC-Hib
Description: Safety was assessed as the number of subjects who reported solicited local reactions from day 1 through day 7 after each vaccination of MenC-CRM administered at 2 months (vaccination 1) and 5 months (vaccination 2). MenC-Hib was administered at 12 months of age (vaccination 3).
Time Frame: Day 1 through day 7 after each vaccination
Population: Analysis was performed on the safety set.
Measure: Number; unit: Number of subjects
Arm/Group | rMenB | rMenB+OMV | Routine | Routine+OMV
Number analyzed (Participants) | 48 | 49 | 25 | 24
Number of subjects
  Tenderness - Vaccination 1 | 7 | 8 | 7 | 5
  Tenderness - Vaccination 2 (N=48,48,25,24) | 7 | 10 | 3 | 6
  Tenderness - Vaccination 3 (N=45,48,24,23) | 8 | 15 | 5 | 5
  Erythema - Vaccination 1 | 37 | 44 | 24 | 21
  Erythema - Vaccination 2 (N=48,48,25,24) | 42 | 43 | 21 | 21
  Erythema - Vaccination 3 (N=45,48,24,23) | 44 | 45 | 22 | 23
  Induration - Vaccination 1 | 12 | 16 | 10 | 7
  Induration - Vaccination 2 (N=48,48,25,24) | 13 | 21 | 11 | 11
  Induration - Vaccination 3 (N=45,48,24,23) | 21 | 24 | 12 | 16

12. Primary Outcome: Number of Subjects Who Reported Solicited Systemic Reactions And Other Indicator of Reactogenicity After Each Vaccination Administered During Study
Description: Safety was assessed as the number of subjects who reported solicited systemic reactions and other indicator of reactogenicity from day 1 through day 7 after each vaccination administered during study as follow: rMenB vaccine with and without OMV, PC7, DTaP-Hib-IPV at 2 months (vaccination 1), MenC-CRM, DTaP-Hib-IPV at 3 months (vaccination 2), rMenB vaccine with and without OMV, PC7, DTaP-Hib-IPV at 4 months (vaccination 3), MenC-CRM at 5 months (vaccination 4), rMenB vaccine with and without OMV at 6 months (vaccination 5; rMenB and rMenB+OMV groups only), rMenB vaccine with and without OMV at 12 months (vaccination 5; routine and routine+OMV groups only), and rMenB vaccine with and without OMV (vaccination 6; rMenB and rMenB+OMV groups only).
Time Frame: Day 1 through day 7 after each vaccination
Population: Analysis was performed on the safety set.
Measure: Number; unit: Number of subjects
Arm/Group | rMenB | rMenB+OMV | Routine | Routine+OMV
Number analyzed (Participants) | 48 | 50 | 25 | 24
Number of subjects
  Change in eating habits - Vaccination 1 | 7 | 13 | 11 | 5
  Change in eating habits- Vaccin 2 (N=48,49,25,24) | 4 | 6 | 3 | 1
  Change in eating habits- Vaccin 3 (N=48,48,25,24) | 12 | 9 | 3 | 4
  Change in eating habits- Vaccin 4 (N=48,48,25,24) | 3 | 3 | 1 | 1
  Change in eating habits- Vaccin 5 (N=47,48,24,23) | 7 | 14 | 6 | 6
  Change in eating habits- Vaccin 6 (N=45,48,25,24) | 11 | 13 | 0 | 0
  Sleepiness - Vaccination 1 | 32 | 32 | 19 | 15
  Sleepiness - Vaccination 2 (N=48,49,25,24) | 19 | 17 | 12 | 9
  Sleepiness - Vaccination 3 (N=48,48,25,24) | 15 | 21 | 6 | 7
  Sleepiness - Vaccination 4 (N=48,48,25,24) | 5 | 7 | 6 | 3
  Sleepiness - Vaccination 5 (N=47,48,24,23) | 5 | 20 | 5 | 10
  Sleepiness - Vaccination 6 (N=45,48,25,24) | 4 | 13 | 0 | 0
  Vomiting - Vaccination 1 | 9 | 3 | 7 | 5
  Vomiting - Vaccination 2 (N=48,49,25,24) | 4 | 1 | 5 | 2
  Vomiting - Vaccination 3 (N=48,48,25,24) | 3 | 5 | 1 | 1
  Vomiting - Vaccination 4 (N=48,48,25,24) | 3 | 1 | 1 | 2
  Vomiting - Vaccination 5 (N=47,48,24,23) | 6 | 5 | 1 | 3
  Vomiting - Vaccination 6 (N=45,48,25,24) | 4 | 3 | 0 | 0
  Diarrhea - Vaccination 1 | 13 | 5 | 4 | 7
  Diarrhea - Vaccination 2 (N=48,49,25,24) | 7 | 5 | 4 | 3
  Diarrhea - Vaccination 3 (N=48,48,25,24) | 8 | 5 | 3 | 4
  Diarrhea - Vaccination 4 (N=48,48,25,24) | 5 | 2 | 3 | 3
  Diarrhea - Vaccination 5 (N=47,48,24,23) | 1 | 4 | 1 | 1
  Diarrhea - Vaccination 6 (N=45,48,25,24) | 7 | 5 | 0 | 0
  Irritability - Vaccination 1 | 34 | 37 | 17 | 15
  Irritability - Vaccination 2 (N=48,49,25,24) | 26 | 29 | 14 | 13
  Irritability - Vaccination 3 (N=48,48,25,24) | 27 | 34 | 13 | 12
  Irritability - Vaccination 4 (N=48,48,25,24) | 15 | 15 | 7 | 6
  Irritability - Vaccination 5 (N=47,48,24,23) | 17 | 30 | 10 | 13
  Irritability - Vaccination 6 (N=45,48,25,24) | 20 | 30 | 0 | 0
  Unusual crying - Vaccination 1 | 11 | 9 | 8 | 7
  Unusual crying - Vaccination 2 (N=48,49,25,24) | 7 | 6 | 5 | 1
  Unusual crying - Vaccination 3 (N=48,48,25,24) | 11 | 7 | 9 | 6
  Unusual crying - Vaccination 4 (N=48,48,25,24) | 5 | 3 | 3 | 2
  Unusual crying - Vaccination 5 (N=47,48,24,23) | 3 | 10 | 3 | 4
  Unusual crying - Vaccination 6 (N=45,48,25,24) | 3 | 5 | 0 | 0
  Rash - Vaccination 1 (N=48,50,25,24) | 10 | 2 | 2 | 3
  Rash - Vaccination 2 (N=48,49,25,24) | 6 | 3 | 3 | 2
  Rash - Vaccination 3 (N=48,48,25,24) | 7 | 5 | 0 | 2
  Rash - Vaccination 4 (N=48,48,25,24) | 9 | 4 | 3 | 4
  Rash - Vaccination 5 (N=47,48,24,23) | 7 | 7 | 5 | 1
  Rash - Vaccination 6 (N=45,48,25,24) | 6 | 8 | 0 | 0
  Fever (≥38 °C) - Vaccination 1 (N=48,50,25,23) | 1 | 9 | 0 | 1
  Fever (≥38 °C) - Vaccination 2 (N=48,49,25,24) | 0 | 0 | 1 | 1
  Fever (≥38 °C) - Vaccination 3 (N=48,48,25,24) | 3 | 4 | 2 | 0
  Fever (≥38 °C) - Vaccination 4 (N=48,48,25,24) | 3 | 0 | 2 | 1
  Fever (≥38 °C) - Vaccination 5 (N=47,48,24,23) | 1 | 2 | 4 | 4
  Fever (≥38 °C) - Vaccination 6 (N=45,48,25,24) | 3 | 3 | 0 | 0
  Analgesic/Antipyretic Med. Used-Vaccination 1 | 15 | 29 | 10 | 8
  Analg. Antipyr. Med. Used-Vaccin 2 (N=48,49,25,24) | 15 | 23 | 10 | 8
  Analg. Antipyr. Med. Used-Vaccin 3 (N=48,48,25,24) | 23 | 31 | 14 | 10
  Analg. Antipyr. Med. Used-Vaccin 4 (N=48,48,25,24) | 10 | 17 | 3 | 9
  Analg. Antipyr. Med. Used-Vaccin 5 (N=47,48,24,23) | 15 | 30 | 9 | 13
  Analg. Antipyr. Med. Used-Vaccin 6 (N=45,48,25,24) | 16 | 33 | 0 | 0

13. Primary Outcome: Percentage of Subjects With Fourfold Rises in Bactericidal Titers Against Meningococcal Strains One Month After Third-Dose of Infants Series Vaccination or rMenB Vaccine With and Without OMV-NZ.
Description: Percentage of subjects fourfold increase in bactericidal titers against meningococcal strains 44/76-SL, 5/99 and NZ98/254 were measured at one month after third-dose and calculated respect to baseline titers.
Time Frame: 30 days after the third vaccination
Population: Analysis was performed on the Per Protocol Set (PP) set, i.e. all subjects in the enrolled population who received all the relevant doses of vaccine correctly; provided evaluable serum samples at the relevant time points, and had no major protocol violation as defined prior to analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 37 | 40
Percentage of Subjects
  Str. 44/76-SL 4-fold Rise-Post-3rd dose (N=36,39) | 69 [52 to 84] | 85 [69 to 94]
  Str. 5/99-SL 4-fold Rise-Post-3rd dose (N=32,37) | 97 [84 to 100] | 92 [78 to 98]
  Str. NZ98/254-4-fold Rise-Post-3rd dose (N=37,40) | 3 [0.068 to 14] | 78 [62 to 89]

14. Primary Outcome: Geometric Mean Ratios to Baseline Against a Panel of Genetically Distinct Meningococcal Strains 30 Days After the Third Immunization.
Description: Geometric Mean Ratios (GMRs) as measure of the bactericidal activity against the for the three major meningococcal B strains (Strain 44/76-SL, Strain 5/99, Strain NZ98/254) in subjects treated with Novartis rMenB Vaccine +/- OMV NZ (Groups I and II) at 30 days after the third immunization. The analysis was done on the Per Protocol population at one month after third injection.
Time Frame: At baseline (pre-vaccination) and 30 days after the third vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 37 | 40
Ratio
  Strain 44/76-SL (1 Month After 3rd | 9.89 [5.79 to 17] | 21 [13 to 34]
  Strain 5/99 (1 Month After 3rd Vacc; | 131 [78 to 220] | 91 [53 to 158]
  Strain NZ98/254 (1 Month After 3rd | 0.91 [0.67 to 1.25] | 16 [9.2 to 28]

15. Secondary Outcome: Geometric Mean Ratios to Baseline Against a Panel of Genetically Distinct Meningococcal Strains 30 Days After a Single Dose Administered at 12 Months of Age
Description: Geometric Mean Ratios to baseline against a panel of genetically distinct meningococcal strains 30 days after a single dose administered at 12 months of age.
Time Frame: 1 month after first vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Routine | Routine+OMV
Number analyzed (Participants) | 22 | 22
Ratio
  44/76-SL (1 month after first Vacc; N=22, 22) | 1.51 [1.02 to 2.22] | 3.21 [1.9 to 5.41]
  5/99 (1 month after first Vacc; N=21, 22) | 73 [53 to 101] | 8 [4.2 to 15]
  NZ98/254 (1 month after first Vacc; N=21, 22) | 0.97 [0.9 to 1.04] | 1.66 [1.12 to 2.45]

16. Secondary Outcome: Percentages of Subjects With Fourfold Rises in Bactericidal Titers After the Second Immunization and at 12 Months Age
Description: Percentages of subjects treated with Novartis rMenB Vaccine +/- OMV NZ (Groups I and II) with fourfold rises in bactericidal titers for the three meningococcal B strains (Strain 44/76-SL, Strain 5/99, Strain NZ98/254) at 30 days after the second vaccination and at 12 months age, i.e. 6 months after third (pre-booster) vaccination, and 1 month after fourth (booster) vaccination. The analysis was done on the Per Protocol population 30 days after the second vaccination and at 12 months age.
Time Frame: At pre-vaccination and 30 days post the 2nd vaccination and at 12 months age, and 1 month post 4th (booster) vaccination.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 41 | 44
Percentages of Subjects
  Strain 44/76-SL (1 Month After 2nd Vacc; N=40, 37) | 50 [34 to 66] | 86 [71 to 95]
  Strain 5/99 (1 Month After 2nd Vacc; N=36, 33) | 89 [74 to 97] | 94 [80 to 99]
  Strain NZ98/254 (1 Month After 2nd Vacc N=41, 38) | 2 [0.062 to 13] | 55 [38 to 71]
  44/76-SL (6 months after pre-booster; N=40, 44) | 45 [29 to 62] | 41 [26 to 57]
  5/99 (6 months after pre-booster; N=37, 40) | 84 [68 to 94] | 65 [48 to 79]
  NZ98/254 (6 months after pre-booster; N=41, 44) | 2 [0.062 to 13] | 23 [11 to 38]
  44/76-SL (1 month after 4th (booster); N=37, 30) | 92 [78 to 98] | 93 [78 to 99]
  5/99 (1 month after 4th (booster); N=33, 27) | 95 [85 to 100] | 97 [83 to 100]
  NZ98/254 (1 month after 4th (booster); N=38, 29) | 0 [0 to 9] | 76 [56 to 90]

17. Secondary Outcome: Percentages of Subjects With Bactericidal Titers, BCA, ≥1:4 After the Second Immunization and at 12 Months Age
Description: Percentages of subjects treated with Novartis rMenB Vaccine +/- OMV NZ (Groups I and II) with a BCA titer ≥1:4 for the three meningococcal B strains (Strain 44/76-SL, Strain 5/99, Strain NZ98/254) at 30 days after the second vaccination and at 12 months age, and 1 month after fourth (booster) vaccination. The analysis was done on the Per Protocol population.
Time Frame: At baseline (pre-vaccination) and 30 days after the second vaccination and at 12 months age.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 46 | 46
Percentages of Subjects
  Strain 44/76-SL (Pre-Vaccination; N=45, 45) | 11 [4 to 24] | 11 [4 to 24]
  Strain 5/99 (Pre-vaccination; N=42, 43) | 7 [1 to 19] | 14 [5 to 28]
  Strain NZ98/254 Pre-Vaccination; N=46, 46) | 4 [1 to 15] | 9 [2 to 11]
  Strain 44/76-SL (1 Month After 2nd Vacc; N=40, 37) | 58 [41 to 73] | 95 [82 to 99]
  Strain 5/99 (1 Month After 2nd Vacc; N=36, 33) | 89 [74 to 97] | 100 [89 to 100]
  Strain NZ98/254 (1 Month After 2nd Vacc; N=41, 38 | 5 [1 to 17] | 74 [57 to 87]
  44/76-SL (6 months after pre-booster; N=40, 44) | 70 [53 to 83] | 68 [52 to 81]
  Strain 5/99 (6 months after prebooster; N=37, 40) | 92 [78 to 98] | 88 [73 to 96]
  NZ98/254 (6 months after pre-booster; N=41, 44) | 5 [1 to 17] | 36 [22 to 52]
  44/76-SL (1 month after booster; N=38, 31) | 100 [91 to 100] | 100 [89 to 100]
  5/99 (1 month after booster; N=34, 30) | 97 [85 to 100] | 97 [83 to 100]
  NZ98/254 (1 month after booster; N=39, 31) | 3 [0.065 to 13] | 94 [79 to 99]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected throughout the study (day 1 through 481).
Description: >5% Adverse Events (AEs) included the solicited local and systemic reactions collected from day 1 through day 7 after each vaccination, and non-serious unsolicited AEs collected from day 8 through day 30 after each vaccination.
Arm/Group | rMenB | rMenB+OMV | Routine | Routine+OMV
Serious Adverse Events (participants affected / at risk) | 3/48 | 9/50 | 4/25 | 2/24
Other Adverse Events (participants affected / at risk) | 48/48 | 50/50 | 25/25 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rMenB (N=48) | rMenB+OMV (N=50) | Routine (N=25) | Routine+OMV (N=24)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rMenB (N=48) | rMenB+OMV (N=50) | Routine (N=25) | Routine+OMV (N=24)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 10 (13) | 4 (4) | 5 (7)
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (7) | 1 (2) | 1 (1)
Somnolence (Nervous system disorders) | 37 (97) | 40 (127) | 22 (52) | 20 (48)
Crying (General disorders) | 26 (51) | 24 (49) | 15 (33) | 12 (21)
Injection Site Bruising (General disorders) | 4 (4) | 4 (5) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 47 (499) | 49 (532) | 25 (211) | 24 (199)
Injection site induration (General disorders) | 41 (218) | 45 (50) | 22 (99) | 24 (130)
Injection Site pain (General disorders) | 36 (145) | 37 (181) | 13 (50) | 18 (64)
Pyrexia (General disorders) | 11 (15) | 15 (20) | 6 (12) | 6 (8)
Vaccination Site Erythema (General disorders) | 3 (5) | 4 (7) | 2 (2) | 2 (3)
Irritability (Psychiatric disorders) | 42 (170) | 48 (222) | 23 (84) | 24 (81)
Eating disorder (Psychiatric disorders) | 27 (52) | 32 (72) | 15 (35) | 12 (20)
Diarrhoea (Gastrointestinal disorders) | 26 (53) | 22 (32) | 13 (24) | 12 (29)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 2 (2)
Teething (Gastrointestinal disorders) | 11 (17) | 15 (20) | 3 (3) | 5 (6)
Vomiting (Gastrointestinal disorders) | 22 (36) | 16 (24) | 12 (23) | 12 (17)
Eczema (Skin and subcutaneous tissue disorders) | 8 (9) | 6 (6) | 2 (2) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 20 (60) | 19 (36) | 10 (17) | 7 (14)
Bronchiolitis (Infections and infestations) | 7 (9) | 2 (3) | 1 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 8 (13) | 5 (5) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (3) | 4 (4) | 2 (2) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gastroenteritis Viral (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Otitis Media (Infections and infestations) | 6 (6) | 7 (7) | 3 (4) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 5 (5) | 12 (16) | 2 (5) | 5 (6)
Upper Respiratory Tract Infection (Infections and infestations) | 10 (10) | 12 (13) | 3 (4) | 2 (2)
Rhinitis (Infections and infestations) | 19 (29) | 19 (25) | 4 (5) | 7 (9)
Varicella (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (4)
Viral Rash (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (2) | 3 (3) | 0 (0)
Vaccination Site Induration (General disorders) | 5 (9) | 6 (8) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days